CLINICAL TRIAL: NCT06781450
Title: Retrospective Observational Study in Patients With Relapsed / Refractory Primary Mediastinal Lymphoma Treated With Pembrolizumab or Nivolumab in Combination With Brentuximab Vedotin in a Real-life Context
Brief Title: Study in Patients With Relapsed/Refractory Primary Mediastinal Lymphoma Treated With Pembrolizumab or Nivolumab in Combination With Brentuximab Vedotin in a Real-life Context
Acronym: PRIMICI
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PRIMICI
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-10

CONDITIONS: Primary Mediastinal B Cell Lymphoma
Keywords: pembrolizumab; nivolumab; brentuximab vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational, Non-Interventional, Retrospective, Multicenter Study Focusing on the Efficacy and Safety of Pembrolizumab Monotherapy and Nivolumab in Combination With Brentuximab Vedotin in Clinical Practice Patients With Primary Mediastinal B Cell Lymphoma Relapsed/Refractory

DETAILED DESCRIPTION:
Observational, non-interventional, retrospective, multicentre study focusing on the efficacy and safety of pembrolizumab as monotherapy and nivolumab in combination with brentuximab vedotin in daily clinical practice in patients with Primary Mediastinal B Cell Lymphoma Relapsed/Refractory. The study aims to retrospectively evaluate the efficacy in terms of overall response rate (ORR, sum of complete response rate [CR] and partial response rate [PR]) of pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin in patients with Primary Mediastinal B Cell Lymphoma Relapsed/RefractoryL treated in a real-life setting from November 2020 until November 2021.

Secondary objectives

* To assess efficacy, in terms of:
* Duration of response (DoR)
* Progression-free survival (PFS)
* Overall survival (OS)
* Disease-free survival (DFS)
* Best response rate (achieved at any time during treatment)
* To evaluate the safety and tolerability of pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin The study will include patients with Primary Mediastinal B Cell Lymphoma Relapsed/Refractory treated with pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin in a real-life setting from November 2020 until November 2021.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of Primary Mediastinal B Cell Lymphoma Relapsed/Refractory patients who underwent pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin in a real-life context with till Novembre 2021
2. Age ≥ 18 years at enrollment
3. Signature of written informed consent (where applicable)

Exclusion Criteria:

1. Primary Mediastinal B Cell Lymphoma Relapsed/Refractory patients who underwent pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin in a clinical trial context.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Primary Mediastinal B Cell Lymphoma Relapsed/Refractory treated with pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin in a real-life context with till Novembre 2021
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | at the end of treatment, through study completion, an average of 2 years
  The study aims to retrospectively evaluate the efficacy in terms of overall response rate (ORR, the sum of complete response [CR] and partial response [PR] rate) of pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin in patients with Primary Mediastinal B Cell Lymphoma Relapsed/Refractory treated in a real-life setting from November 2020 through November 2021

SECONDARY OUTCOMES:
Duration of Response (DoR) | through study completion, an average of 2 years
  Duration of Response (DoR)
Progression Free Survival (PFS) | through study completion, an average of 2 years
  Progression Free Survival (PFS)
Overall Survival (OS) | through study completion, an average of 2 years
  Overall Survival (OS)
Disease Free Survival (DFS) | through study completion, an average of 2 years
  Disease Free Survival (DFS)
Best response rate (BRR) | through study completion, an average of 2 years
  Best response rate (BRR)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 2 years
  safety and tolerability of pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin
Incidence of Treatment-Emergent Serious Adverse Events [Safety and Tolerability] | through study completion, an average of 2 years
  safety and tolerability of pembrolizumab as a single agent and nivolumab in combination with brentuximab vedotin

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna
  - Azienda Ospedaliera Universitaria- POLICLINICO BARI, Bari
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan

IPD SHARING:
Plan to Share IPD: No